CLINICAL TRIAL: NCT05865743
Title: PERi-operative Selective Decontamination of the Digestive Tract to Prevent Severe Infectious Complications After Esophagectomy: a Randomized Multicenter Clinical Trial in Patients with Primary Resectable Esophageal Carcinoma (cT1-4, N0-3, M0)
Brief Title: Perioperative SDD to Prevent Infectious Complications After Esophagectomy
Acronym: PERSuaDER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-504144-33-00
Record Dates: First submitted 2023-04-25; First posted 2023-05-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SDD treatment (Experimental): Standard of care + SDD treatment
  Interventions: Drug: SDD
- Standard of care (No Intervention): Standard of care

INTERVENTIONS:
Drug: SDD — The intervention group receives SDD treatment additional to standard care, comprising two distinct liquids for oral administration: first the 5 ml amphotericin B suspension (100 mg/ml) and subsequently the 5 ml "SDD base for suspension", containing both colistin sulphate (20 mg/ml) and tobramycin sulphate (16 mg/ml).
  Patients take the 5 ml amphotericin B, followed by the 5 ml "SDD base for suspension", four times daily for one week, starting three days prior to the surgery. On the day of surgery, intake is limited to an early morning and a late evening dose.
  Other Names: Standard of care
  Arms: SDD treatment

SUMMARY:
The primary aim of the PERSuaDER-trial is to evaluate the effect of SDD on infectious complications after esophagectomy, focussed on the prevention of pneumonia

DETAILED DESCRIPTION:
Esophagectomy is a complex surgical procedure, associated with significant morbidity and mortality rates. Most postoperative complications are caused by infections (10-30%). These are thought to arise from (micro-)aspiration of bacteria residing in the oropharyngeal and gastrointestinal (GI) tract, leading to (respiratory) infections. Selective decontamination of the digestive tract (SDD) is a prophylactic antibiotic strategy that aims to prevent postoperative infections. Pathogenic aerobic gram-negative rods and yeasts tract are reduced, while anaerobic, protective microbiota are preserved. SDD has been shown to lower the risk for respiratory infections in an intensive care setting. Establishing SDD as effective addition to the standard care of esophagectomy patients is expected to increase their chance of survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary esophageal adenocarcinoma or squamous cell carcinoma (cT1b-4a,N0-3,M0) in the mid or distal esophagus or at the level of the gastro-esophageal junction scheduled for undergoing transthoracic esophagectomy with curative intent or for esophageal reconstruction with a gastric or jejunal interposition
* Age ≥ 18 years,
* Able to give written informed consent.

Exclusion Criteria:

* Patients planned for rescue surgery,
* Patients planned for colonic interposition,
* Known or suspected pregnancy,
* Patients who have undergone upper GI surgery within 30 days before randomization,
* Unable to understand the study information, study instructions and give informed consent.
* Patients enrolled in a trial that would interact with the intervention
* Patients with a known allergy, sensitivity, or interaction to investigational medicinal product.
* Patients with known/documented colonization of Enterobacteriaceae and or Pseudomonas Aeruginosa that are resistant to both tobramycin/gentamicin and to carbapenem antibiotics
* Patients undergoing CVVH.
* Patients with documented chronic renal failure (GFR < 15 mls/min) or who are on chronic intermittent hemo- or peritoneal dialysis,
* Women of childbearing potential at risk of pregnancy, not using adequate contraception,
* Patients with the inability to swallow the SDD
* Patients with pre-existing degenerative neuromuscular diseases like, but not limited to, myasthenia gravis or Parkinson disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 854 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
the cumulative incidence of postoperative pneumonia within 30 days after surgery | Within 30 days after surgery
  The primary outcome parameter is the cumulative incidence of postoperative pneumonia within 30 days after surgery. Pneumonia will be defined by the following criteria:
  * Positive sputum culture OR
  * Presence of a new progressive radiographic infiltrate plus at least 2 of the following clinical features:
  * Fever > 38.5°C
  * Leukocytosis (>11.0) or leukopenia (<4.0)
  * Purulent secretions

SECONDARY OUTCOMES:
the cumulative incidence of all postoperative infectious complications within 30 days after surgery | Within 30 days after surgery
  the cumulative incidence of all postoperative infectious complications as registered in DUCA (postoperative pneumonia, urinary tract infection, wound infection/abscess requiring wound opening or antibiotic treatment, central line infection requiring line removal or antibiotic treatment, intra-thoracic/intra-abdominal abscess, generalised sepsis as defined by Evans, Rhodes (2), infections with Highly-resistant Enterobacteriaceae (HRE) and Clostridium difficile, other infections requiring antibiotics. All these complications are then graded according to the Clavien-Dindo classification
the cumulative incidence of anastomotic leakage within 30 days after esophagectomy for which endoscopic, radiologic, or surgical re-intervention is needed | Within 30 days after surgery
  the cumulative incidence of anastomotic leakage within 30 days after esophagectomy for which endoscopic, radiologic, or surgical re-intervention is needed. This corresponds to the definition of the ECCG of anastomotic leakage type II and III Low, Alderson (3). Anastomotic leakage is defined by contrast leakage on CT-scan with intravenous and oral contrast (swallow CT-scan) upon clinical suspicion, by endoscopy or by drainage of ingested materials into the chest tube (thoracic anastomoses) or ingested materials or saliva into cervical wound (cervical anastomosis) or signs of anastomotic leakage during re-intervention or autopsy
the mortality rate within 90 days after surgery | Within 90 days after surgery
  All-cause mortality
the rate of re-operation within 30 days after surgery | Within 30 days after surgery
  Rate of re-operation
the postoperative length of stay on the intensive care unit (ICU) within 6 months after surgery defined in days | Within 6 months after surgery
  the postoperative length of stay on the intensive care unit (ICU), including re-admissions
the postoperative length of the total hospital stay within 6 months after surgery defined in days | Within 6 months after surgery
  the postoperative length of the total hospital stay, including re-admissions for any reasons within 6 months after surgery
Quality of life questionnaire (EORTC QLQ C30) | After 30 days, 3 months and 6 months after surgery
  This study aims to determine the differences in the quality of life after 30 days, 3 months and 6 months after surgery using the following questionnaire European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC QLQ C30): All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Using paper or electronical forms, whatever a participant prefers paper forms or a printed version will be provided.
Quality of life questionnaire (EORTC QLQ OG25) | After 30 days, 3 months and 6 months after surgery
  This study aims to determine the differences in the quality of life after 30 days, 3 months and 6 months after surgery using the following questionnaire European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Oesophago Gastric module 25 (EORTC QLQ OG25): All of the scales and single-item measures range in score from 0 to 100. A high score for all the scales and single-items represents a high level of symptomatology or problems. Using paper or electronical forms, whatever a participant prefers paper forms or a printed version will be provided.
Quality of life questionnaire (EQ-5D-5L) | After 30 days, 3 months and 6 months after surgery
  •This study aims to determine the differences in the quality of life after 30 days, 3 months and 6 months after surgery using the following questionnaire The 5-level EuroQol-5D-5L (EQ-5D-5L). This descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. It is scaled from 0 to 100%. A higher score indicates a higher quality of life. Using paper or electronical forms, whatever a participant prefers paper forms or a printed version will be provided.
Direct and indirect costs defined in Euros | Up to 6 months after surgery
  The in-hospital and societal costs up to 6 months after surgery will be estimated with the help of the medical consumption questionnaire and the productivity cost questionnaire, developed by the iMTA. For Belgium a database cross linkage with the RIZIV/INAMI expenses is foreseen based on data pseudonymized by a Trusted Third Party and handled by KCE. The Belgian national patient identifier number will be used for data linkage with the expenses database of the health insurance provider, but will be withdrawn from the dataset by KCE before the analysis is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Camiel Rosman, Prof, Principal Investigator — RadoudUMC
Locations (2):
- UZ Leuven, Leuven, Belgium
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
A subset of the final data will be made available after an embargo period upon request. Most likely aggregated and filtered in order to maintain anonymity of individual patient data. The choice of online repository still has to be made.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: six months after database lock
Access Criteria: Upon request to the Principal investigator, with a sufficiently substantiated study protocol.

REFERENCES:
- [Background] Low DE, Alderson D, Cecconello I, Chang AC, Darling GE, D'Journo XB, Griffin SM, Holscher AH, Hofstetter WL, Jobe BA, Kitagawa Y, Kucharczuk JC, Law SY, Lerut TE, Maynard N, Pera M, Peters JH, Pramesh CS, Reynolds JV, Smithers BM, van Lanschot JJ. International Consensus on Standardization of Data Collection for Complications Associated With Esophagectomy: Esophagectomy Complications Consensus Group (ECCG). Ann Surg. 2015 Aug;262(2):286-94. doi: 10.1097/SLA.0000000000001098. PMID 25607756
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Derived] Grootenhuis JGA, Seurs W, Garms LM, de Vries M, Ubels S, van Werkhoven HC, Rosman C, Schouten JA, Klarenbeek BR, Van Veer H. PERi-operative Selective Decontamination of the digestive tract to prevent severe infectious complications after Esophageal Resection: study protocol of the PERSuaDER-trial, a multicenter randomized controlled trial in patients with primary resectable esophageal carcinoma. Trials. 2025 Dec 4;27(1):16. doi: 10.1186/s13063-025-09311-w. PMID 41345690
- See also: DUCA Data — https://dica.nl/registratie/maag-en-slokdarmkanker-duca/